CLINICAL TRIAL: NCT02085746
Title: Defining Sexual Activity: How Demographics May Impact Our Definition
Brief Title: Defining Sexual Activity
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Kristie Greene, Female Pelvic Medicine and Reconstructive Surgery PGY7, University of South Florida
Other Study IDs: Pro00015065
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Demographics Effecting One's Definition of Being Sexually Active

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Defining Sexual Activity Questionnaire

SUMMARY:
This will be a descriptive study using patients from the Urogynecology and Urology University of South Florida Clinics and Urology clinic at Tampa General Hospital Healthpark on 30th Street to analyze the impact of demographics on the definition of being sexually active. It is believed one's demographics influence their definition of being sexually active.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women >18 who seek urogynecological/urological treatment
* English speaking
* Willing and able to provide written and informed consent

Exclusion Criteria:

* Men and Women <18
* Not a patient at the appropriate Urogynecological and Urology clinics
* Non-English speaking
* Unable or unwilling to provide written and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female patient over 18 years of age seeking urogynecological/urological treatment at one of the participating clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Definition of Sexual Activity | 6 months
  Based on questionnaire answers, the goal is to define sexual activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Greene, M.D., Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - Tampa General Hospital HealthPark/30th Street, Tampa, Florida
  - University of South Florida Urogynecology Clinic, Tampa, Florida
  - University South Florida Urology Clinic, Tampa, Florida

REFERENCES:
- [Background] Dalpiaz O, Kerschbaumer A, Mitterberger M, Pinggera GM, Colleselli D, Bartsch G, Strasser H. Female sexual dysfunction: a new urogynaecological research field. BJU Int. 2008 Mar;101(6):717-21. doi: 10.1111/j.1464-410X.2007.07442.x. Epub 2008 Jan 10. PMID 18190620
- [Background] Fashokun TB, Harvie HS, Schimpf MO, Olivera CK, Epstein LB, Jean-Michel M, Rooney KE, Balgobin S, Ibeanu OA, Gala RB, Rogers RG; Society of Gynecologic Surgeons' Fellows' Pelvic Research Network. Sexual activity and function in women with and without pelvic floor disorders. Int Urogynecol J. 2013 Jan;24(1):91-7. doi: 10.1007/s00192-012-1848-2. Epub 2012 Jun 29. PMID 22744621
- [Background] Rogers RG, Rockwood TH, Constantine ML, Thakar R, Kammerer-Doak DN, Pauls RN, Parekh M, Ridgeway B, Jha S, Pitkin J, Reid F, Sutherland SE, Lukacz ES, Domoney C, Sand P, Davila GW, Espuna Pons ME. A new measure of sexual function in women with pelvic floor disorders (PFD): the Pelvic Organ Prolapse/Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR). Int Urogynecol J. 2013 Jul;24(7):1091-103. doi: 10.1007/s00192-012-2020-8. Epub 2013 Apr 30. PMID 23632798
- [Background] Tok EC, Yasa O, Ertunc D, Savas A, Durukan H, Kanik A. The effect of pelvic organ prolapse on sexual function in a general cohort of women. J Sex Med. 2010 Dec;7(12):3957-62. doi: 10.1111/j.1743-6109.2010.01940.x. PMID 20646180